CLINICAL TRIAL: NCT04827771
Title: Different Actors for the Same Play: the Impact of the Biologist Performing the Embryo Transfer on the Cycle Outcome
Brief Title: The Impact of the Biologist Performing the Embryo Transfer on the Cycle Outcome
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-407
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective single center analysis which includes all the fresh, IOC (insemination of in vitro matured oocytes) and frozen embryo transfer (ET) performed between January 2000 and December 2019 at Humanitas Fertility Center after IVF-ICSI (In Vitro Fertilization - Intracytoplasmic Sperm Injection) cycles.

The primary objective is to determine the impact of the biologist performing the embryo transfer on the pregnancy probability, in terms of ongoing pregnancy rate (OPR), defined as the number of viable pregnancies that had completed at least 12 weeks of gestation on the total number of ET performed.

Secondary end point is to evaluate whether the biologists improve their performances as their experience increases, allowing the drawing of an ET learning curve in term of pregnancies for the different biologists.

The biologist's experience was assessed in terms of number of previous interventions performed prior to the day of ET. A total of 28 operators were eligible to participate in the study. Any biologists who performed less than 100 ETs was excluded from the analysis.

ELIGIBILITY:
Inclusion criteria:

Exclusion Criteria:

Any biologist who performed less than 100 embryo transfers was excluded from the analysis.

Ages: 18 Years to 43 Years | Sex: Female
Age Groups: Adult
Study Population: All the fresh, IOC (insemination of in vitro matured oocytes) and frozen embryo transfer performed between January 2000 and December 2019 at Humanitas Fertility Center.
  A total of 28 biologist operators were eligible to participate in the study.
Sampling Method: Probability Sample
Enrollment: 30000 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 20 years
  The number of viable pregnancies that had completed at least 12 weeks of gestation per total ETs

REFERENCES:
- [Background] Li H, Li L, Lu X, Sun X, Ng EHY. Comparison of the effect of immediate versus delayed transfer following a stimulated IVF cycle on the ongoing pregnancy rate of frozen-thawed embryo transfer cycles: a study protocol for a randomised controlled trial. BMJ Open. 2018 May 17;8(5):e020507. doi: 10.1136/bmjopen-2017-020507. PMID 29773699